CLINICAL TRIAL: NCT07323433
Title: Efficacy of a Chitosan Dressing in Pulpotomy of Immature Permanent Teeth:Randomized Clinical Trial
Brief Title: Efficacy of a Chitosan Dressing in Pulpotomy of Immature Permanent Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Salsabil Mohammed Naguib, Specialist at Health Insurance Endodontics , Minia city, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chitosan Dressing
Record Dates: First submitted 2025-11-27; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Hemcon Dressing (Active Comparator): About 13 Participants presented with traumatic or caries exposed upper anterior teeth with immature root and they will be subjected to Application of Hemcon Dressing as A dressing material for hemostasis on pulp stump during pulpotomy of the immature teeth.
  Interventions: Procedure: Chitosan Dressing
- Group of Cotton damped with normal saline (Active Comparator): About 13 Participants presented with traumatic or caries exposed upper anterior teeth with immature root and they will be subjected to Application of cotton damped with normal saline for hemostasis on pulp stump during pulpotomy of the immature teeth.
  Interventions: Procedure: Chitosan Dressing

INTERVENTIONS:
Procedure: Chitosan Dressing — To evaluate the effect of chitosan dressing in pulpotomy of immature permanent teeth
  Other Names: Hemcon Dressing; pulpotomy of immature permanent teeth; Cotton damped with normal saline

SUMMARY:
Immature permanent teeth, also known as young permanent teeth, are used to describe teeth with incomplete root formation. Immature permanent teeth are prone to caries and trauma which can cause exposure and degeneration of pulp. Pulp degeneration stops root formation, leaving teeth with open apex. It is vital to preserve the pulp vitality otherwise the incompletion of root might result in the fragility of teeth. Pulpotomy is one of the most widely used methods in preserving vital pulp in teeth, which is of great significance in achieving continue root formation in immature permanent teeth suffering from dental caries or trauma. Pulpotomy is recommended by the American Association of Pediatric Dentistry for the management of pulp exposure in immature permanent teeth to achieve apexogenesis (continued root formation and closure of apex). In this procedure, coronal pulp tissue is removed in order to eliminate the infected or contaminated pulp and to reach the healthy vital pulp followed by coverage with biocompatible material.

DETAILED DESCRIPTION:
Immature permanent teeth, also known as young permanent teeth, are used to describe teeth with incomplete root formation. Immature permanent teeth are prone to caries and trauma which can cause exposure and degeneration of pulp. Pulp degeneration stops root formation, leaving teeth with open apex. It is vital to preserve the pulp vitality otherwise the incompletion of root might result in the fragility of teeth. Pulpotomy is one of the most widely used methods in preserving vital pulp in teeth, which is of great significance in achieving continue root formation in immature permanent teeth suffering from dental caries or trauma. Pulpotomy is recommended by the American Association of Pediatric Dentistry for the management of pulp exposure in immature permanent teeth to achieve apexogenesis (continued root formation and closure of apex). In this procedure, coronal pulp tissue is removed in order to eliminate the infected or contaminated pulp and to reach the healthy vital pulp followed by coverage with biocompatible material.

Clinically, the characteristic and the extent of pulpal hemorrhage at the exposure site are the most important outcome predictors for assessing pulpal status.

reported that excessive bleeding from the pulp revealed a significantly lower incidence of success compared with moderate bleeding. A variety of solutions and methods have been used to obtain pulpal hemostasis. Despite its limited effect on pulpal healing, sterile saline is a frequently used agent. Sodium hypochlorite (NaOCl), in concentrations of 0.5percent, achieves hemostasis without affecting pulpal repair mechanism and healing.

Hemostatic dressings have emerged as valuable adjuncts in dentistry, offering effective and efficient control of bleeding during various dental procedures. The different types of hemostatic dressings, including oxidized cellulose, gelatin- based, chitosan, and calcium-based dressings, provide localized hemostasis, reduce chair time, and improve patient outcomes.

Recently, the concept of lesion sterilization and tissue repair therapy involve the use of a mixture of antibacterial drugs for disinfection. Repair of damaged tissues can be expected if lesions are disinfected.

Chitosan is a natural and non-toxic polysaccharide with unique biological properties such as antimicrobial, anti- fungal, anti-inflammatory, antiseptic, antitumor, hemostatic,

immune adjuvant, regenerative effect and wound healing. In dentistry, it can be used as a dental pulp capping material, mouth rinse, chewing gum, drug device for root canal disinfection, topical treatment of periodontitis and blood hemostasis after tooth extraction.

Chitosan is the most abundant biopolymer on the earth derived from chitin. It shows a remarkable effective broad spectrum antibacterial action attributed to its cationic nature. It interacts with the -ve charged bacterial cell membranes, leading to leakage of the intracellular constituents and ultimately cell death due to increasing the membrane permeability. Also, chitosan possesses a variety of other biological properties as being biodegradable, biocompatible.

ELIGIBILITY:
Inclusion Criteria:

* Patients with immature maxillary anterior teeth.
* Patients with caries or traumatic exposed teeth .
* Patients should be free from any systemic disease that may affect normal healing and predictable outcome class I ASA .
* Patients who will agree to the consent and will commit to follow-up period.

Exclusion Criteria:

* Patients with mature roots.
* Patients with any systemic disease that may affect normal healing.
* Patients with signs of periapical inflammation.
* Patients who could/would not participate in a 1-year follow-up.
* Teeth with periodontal involvement.
* Teeth with vertical root fractures.
* Non- restorable teeth.
* cases with previously initiated endodontic treatment.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Post Operative Pain | 6 Months till 12 months
  Assessment of the post operative pain via Numerical Pain Rating Scale (NRS) where the level of pain will be recorded as follows: 0 reading represents "no pain" ; 1- 3 reading represents "mild pain" ; 4- 6 reading represents "moderate pain" and 7- 10 reading represents "severe pain".

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa Ahmed Ebrahem, Professor, Study Chair — Department of endodontics Dean of Faculty of Dentistry Fayoum University
Locations (1):
- Minia University Hospital, Minya, Egypt